CLINICAL TRIAL: NCT04220554
Title: Long-term Improvement of Psoriasis Patients' Adherence to Topical Drugs: Testing a Patient-supporting Intervention Delivered by Healthcare Professionals
Brief Title: Improvement of Psoriasis Patients' Adherence to Topical Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Tiedemann Svendsen, Specialist in dermato-venereology, MD, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LF-OC-000048
Record Dates: First submitted 2019-12-06; First posted 2020-01-07 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group:
  All participants will be instructed how to use of the medication according to "the fingertip unit for topical steroids". All participants will be prescribed topical drugs based on shared decision between the prescriber and patient. The topical drugs will be either moderate corticosteroids (clobetasone-17-butyrate or hydrocortisone-17-butyrate), potent corticosteroids (betamethasone-17-valerate and betamethasone, mometasone furoate, fluocinolone acetonide or fluocinonide), very potent corticosteroids (clobetasol propionate), corticosteroids with antimicrobials (betamethasone and clioquinol, betamethasone and fusidic acid or fluocinolone acetonide and clioquinol), corticosteroid with calcipotriol or calcipotriol cream.
  During the study period, a nurse or pharmaconomist will deliver;
  * Improved support and instructions to the patients
  * Patients will receive a diary and access to more consultations.
  Interventions: Other: Improved support by health-care professionals
- Non-intervention group (No Intervention): All participants will be instructed how to use of the medication according to "the fingertip unit for topical steroids". All participants will be prescribed topical drugs based on shared decision between the prescriber and patient. The topical drugs will be either moderate corticosteroids (clobetasone-17-butyrate or hydrocortisone-17-butyrate), potent corticosteroids (betamethasone-17-valerate and betamethasone, mometasone furoate, fluocinolone acetonide or fluocinonide), very potent corticosteroids (clobetasol propionate), corticosteroids with antimicrobials (betamethasone and clioquinol, betamethasone and fusidic acid or fluocinolone acetonide and clioquinol), corticosteroid with calcipotriol or calcipotriol cream.

INTERVENTIONS:
Other: Improved support by health-care professionals — Improved support to patients prescribed topical antipsoriatic drugs
  Arms: Intervention group

SUMMARY:
Psoriasis affects 2-4% of the Western adult population and is a socio-economic burden for patients and society. Topical drugs are recommended as first-line treatment for mild-to-moderate psoriasis, but low adherence is a barrier for treatment success. There is a need for improved patient support for psoriasis patients, which is suggested to improve long-term use of topical drugs.

The project aims to test whether a patient-supporting intervention delivered by healthcare professionals can improve the use of topical drugs. The intervention design is based on experiences with previous adherence-improving studies consisting of digital support by conducting a systematic literature search and holding focus groups with patients as well as healthcare professionals. The intervention consists of shared decision-making with patients, nurses and doctors, frequent consultations, easy access to healthcare professionals through video or in-office consultations and holding patients accountable for taking the medication.

The intervention will be tested in a randomized controlled trial: during a 48 week period, a group of patients (18-85 years of age) diagnosed with mild-to-moderate psoriasis and treated with topical drugs will be randomized to an intervention (n=40) or non-intervention group (n=40). The primary outcome will be severity of psoriasis and secondary outcomes primary adherence (i.e., rate of filled prescriptions) and quality of life.

If the intervention can reduce the severity of psoriasis in a significant manner, there is a potential for a national implementation of the intervention.

DETAILED DESCRIPTION:
Background Psoriasis is a chronic inflammatory skin disease affecting 2-4% of the Western adult population. It is associated with many comorbidities, negatively affects quality of life and is a socioeconomic burden for patients and society. Topical drugs are the recommended first-line treatment for mild-to-moderate psoriasis, but adherence rates are low, which is a barrier for treatment success, resulting in a need for systemic or biological treatments, which are associated with more severe adverse events and are more expensive than topical drugs. However, improved adherence to topical drugs is associated with improved efficacy. That is why there is a need for improving psoriasis patients' adherence to topical drugs.

As a supplement to the introduction of new and advanced technology, there is a need for more studies on how to optimize the available healthcare professionals in dermatology clinics. Since dermatologists are a limited resource, there is a need to study how other healthcare professionals, e.g., hospital nurses and pharmaconomists at the pharmacies, can support psoriasis patients in their use of topical drugs.

Hypothesis

A patient-supporting intervention delivered by dermatologists, dermatology nurses and pharmaconomists significantly reduces psoriasis patients' severity of psoriasis compared to standard patient support.

Aims

The aim of the project is to test whether an individualized patient-supporting intervention delivered to psoriasis patients by dermatologists, nurses and pharmaconomists at a dermatology hospital clinic can: 1) reduce the severity of psoriasis, 2) improve quality of life, and 3) improve adherence to prescribed topical drugs.

Ethical considerations

All participants will be fully informed of the purpose of the study, and the study will be performed in accordance with the ethical principles in the Belmont report.

Materials and methods

The study is an investigator-initiated, single-centre, assessor-blinded, parallel group superiority randomized clinical study. Before inclusion of study participants, the study will be approved by the local regional ethics committee.

We will include patients (18-85 years of age) with milder-to-moderate psoriasis.

Outcomes

Outcome measurements will be either patient-reported or assessor-blinded.

Adherence measurements

Primary adherence: Proportion of filled topical prescriptions.

Secondary adherence:

Amount of medication used according to weight of the remains in the used medication packages. Data will be assessed week 48.

Disease severity measurements

Disease severity will be measured by Lattice-System Physician's Global Assessment (LS-PGA) (15), and the quality of life will be measured by the Dermatology Life Quality Index (DLQI). This data will be assessed at baseline, weeks 12, 24, 36 and 48.

Recruitment

Psoriasis patients who use topical treatments and are referred to the Department of Dermatology at Odense University Hospital will be recruited to the project until there is a sufficient number of participants included (n=100).

Hypothesis and expected number of participants

Our null hypothesis is that there is no difference in reduction of psoriasis between the intervention and non-intervention groups.

The sample size was calculated based on data from a previous project with consumption data for the use of prescribed calcipotriol betamethasone dipropionate cutaneous foam over 4 weeks. We expect an 20% difference in the LS-PGA, power 80%, two-sided significance of 95%, allocation of 1: 1 and an expected dropout rate of 25%. When using an unpaired t-test, the calculation resulted in the inclusion of a sample size consisting of 80 participants.

Blinding and randomization

Blinding of the data assessors: When the data assessor obtains baseline data from the study participants, it will be entered by an electronic data collection tool.

Participants will be allocated 1: 1 to an intervention or non-intervention arm via a computer-generated block randomization. The data assessor will be blinded to the allocation.

Statistics

Analysis of the primary outcome: changes in LS-PGA

Changes in LS-PGA measurements from baseline to weeks 12 and from baseline to weeks 24, 36 and 48 will be compared between the two groups by linear mixed model for longitudinal data. LS-PGA will be presented in box plots. As a sensitivity analysis on LS-PGA, the analysis will be carried out excluding missing data and after 100 times multiple imputations by multivariate normal regression on LS-PGA data, without included covariates in addition to with an imputation including treatment, age, sex and smoking as covariates.

Analysis of secondary outcomes: Changes in DLQI and adherence

Changes in DLQI measurements from baseline to weeks 12, 24, 36 and 48 will be compared between the two groups by linear mixed model for longitudinal data. DLQI will be presented in box plots.

For the analysis of adherence (by filled prescriptions, weight and patient reported), we will dichotomize adherence rate with a selected cut-off of 80%, with adherence rates above 80% considered adherent (a cut-off typically used when studying adherence in chronic diseases) [7, 42]. We will compare the dichotomized adherences by using logistic regression.

The statistical analysis will be conducted by an experienced statistician blinded to the intervention. An interim analysis is not planned.

Discussion

This study will demonstrate whether an individualized, optimized patient support delivered by doctors, nurses and pharmaconomists to dermatological patients can optimize the use of topical treatment, reduce the severity of psoriasis and have socioeconomic benefits compared to standard treatment. If the study shows that individualized and optimized patient support is effective, it is intended for the intervention to be implemented in the clinic. In addition, we will work on implementing the intervention nationally by a translational process.

Results from the study may also be referred to other chronic dermatological disorders. The study may be used methodically as a model for additional research projects investigating medical adherence in other chronic skin diseases.

ELIGIBILITY:
Inclusion Criteria: Legally competent patients with milder-to-moderate psoriasis

Exclusion Criteria: Incapable patients not diagnosed with psoriasis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias T Svendsen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Dermatology and Allergy Centre, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Svendsen MT, Feldman SR, Moller S, Kongstad LP, Andersen KE. Long-term improvement of psoriasis patients' adherence to topical drugs: testing a patient-supporting intervention delivered by healthcare professionals. Trials. 2021 Oct 25;22(1):742. doi: 10.1186/s13063-021-05707-6. PMID 34696820
- [Result] Svendsen MT, Feldman SR, Mejldal A, Moller S, Kongstad LP, Andersen KE. Regular support provided by dermatological nurses improves outcomes in patients with psoriasis treated with topical drugs: a randomized controlled trial. Clin Exp Dermatol. 2022 Dec;47(12):2208-2221. doi: 10.1111/ced.15370. Epub 2022 Oct 25. PMID 35973788
- [Result] Svendsen MT, Andersen KE, Feldman SR, Mejldal A, Moller S, Kongstad LP. An effective patient-supporting intervention for topical treatment of psoriasis is also cost-effective. Clin Exp Dermatol. 2023 Oct 25;48(11):1247-1254. doi: 10.1093/ced/llad272. PMID 37585448

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Intervention group:
  All participants will be instructed how to use of the medication according to "the fingertip unit for topical steroids". All participants will be prescribed topical drugs based on shared decision between the prescriber and patient. The topical drugs will be either moderate corticosteroids (clobetasone-17-butyrate or hydrocortisone-17-butyrate), potent corticosteroids (betamethasone-17-valerate and betamethasone, mometasone furoate, fluocinolone acetonide or fluocinonide), very potent corticosteroids (clobetasol propionate), corticosteroids with antimicrobials (betamethasone and clioquinol, betamethasone and fusidic acid or fluocinolone acetonide and clioquinol), corticosteroid with calcipotriol or calcipotriol cream.
  During the study period, a nurse or pharmaconomist will deliver;
  * Improved support and instructions to the patients
  * Patients will receive a diary and access to more consultations.
  Improved support by health-care professionals: Improved support to patients prescribed topical antipsoriatic drugs
Period: Overall Study
Arm/Group | Intervention Group | Non-intervention Group
Started | 51 | 52
Completed | 45 | 47
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Non-intervention Group | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 42 | 80
  >=65 years | 13 | 10 | 23
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 58 [40.0 to 71.0] | 52.5 [42.5 to 66.0] | 55.3 [40.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 51 | 51
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 0 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 51 | 52 | 103
Severity of psoriasis: Lattice System Physician's Global Assessment (LS-PGA) [Mean (Full Range); unit: units on a scale] — Lattice-System Physician's Global Assessment (LS-PGA) (interval scale). From value 1 (no visible psoriasis) to 8 (severely affected by psoriasis)
  units on a scale | 5.3 [2 to 8] | 5.1 [2 to 8] | 5.2 [2 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Severity of Psoriasis
Description: Lattice-System Physician's Global Assessment (LS-PGA) (interval scale). From value 1 (no visible psoriasis) to 8 (severely affected by psoriasis).
Time Frame: Change from baseline at week 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 45 | 47
units on a scale | 2.68 [2.20 to 3.15] | 1.84 [1.46 to 2.22]

2. Secondary Outcome: Secondary Adherence
Description: Proportion of expected consumed amount of topical drugs.
  Secondary adherence was calculated by combining measured amount of medication used (determined by the weight of the remains in the used medication packages) per body surface area unit affected.
  Estimated recommended consumption of medication was 0.5 g per day multiplied by the estimated mean body surface area (BSA) during the whole study period, calculated from BSA measures at baseline and at weeks 12, 24, 36, and 48.
Time Frame: Week 48
Population: The number participants analyzed is not consistent with the participant flow chart, since some patients did not return the medication packages and therefore their data could not be included in the analysis of secondary adherence.
Measure: Mean (95% Confidence Interval); unit: percentage of adherence
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 44 | 44
percentage of adherence | 106 [68 to 144] | 72 [49 to 95]

3. Secondary Outcome: Quality of Life (QOL)
Description: Dermatology Life Quality Index (DLQI) (interval scale). From value 0 (no impact on quality of life) to 30 (severe impact on quality of life).
Time Frame: Change from baseline to week 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Non-intervention Group
Number analyzed (Participants) | 45 | 47
units on a scale | 6.88 [5.83 to 7.93] | 1.55 [0.51 to 2.60]

ADVERSE EVENTS:
Time Frame: 48 weeks.
Description: Adverse event recording was collected by systematic interview and patient charts.
Arm/Group | Intervention Group | Non-intervention Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/52
Serious Adverse Events (participants affected / at risk) | 20/51 | 12/52
Other Adverse Events (participants affected / at risk) | 22/51 | 17/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=51) | Non-intervention Group (N=52)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) — Adverse event lead to hospitalization
Urinary tract infection (Infections and infestations) | 2 (6) | 0 (0) — Adverse event lead to hospitalization
Inflammation of epididymis (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Abscess in anogenital area (Gastrointestinal disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Primary adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Dysregulated diabetes mellitus (Endocrine disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) — Adverse event lead to hospitalization
Mania (Psychiatric disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Adverse event during operation lead to hospitalization
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) — Adverse event lead to hospitalization
Ear stone dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Hepatocellular adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Commotio cerebri (Nervous system disorders) | 0 (0) | 1 (1) — Adverse event lead to hospitalization
Exacerbation of chronic renal failure (Renal and urinary disorders) | 0 (0) | 1 (2) — Adverse event lead to hospitalization
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) — Adverse event lead to hospitalization
Acute sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Adverse event lead to hospitalization
Tongue cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Adverse event lead to hospitalization
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Adverse event lead to hospitalization
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Adverse event lead to hospitalization
Basal cell skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Osteoporosis (Endocrine disorders) | 0 (0) | 1 (1)
Psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=51) | Non-intervention Group (N=52)
Bacterial folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep bacterial inflammation in the subcutaneous tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erysipelas (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Boil (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatophytosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Paronychia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria acuta (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hidrosadenitis suppurativa (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Spontaneous ecchymoses (Skin and subcutaneous tissue disorders) | 10 (10) | 1 (1)
Dysesthesia of the skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Superficial vein trombosis (Vascular disorders) | 0 (0) | 1 (1)
Fractura caput radii (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT04220554/Prot_SAP_000.pdf